CLINICAL TRIAL: NCT04274920
Title: Clinical Response of Human Pulps Capped With Bioactive Glass Incorporated in Resin Composite and Adhesive
Brief Title: Dentin Bridge Formation After Indirect Pulp Capping With Bioactive Glass Incorporated in Resin Composite and Its Adhesive in Comparison With Light Cured Calcium Hydroxide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Heba Arafa Abd El wahab Zahran, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC16-071
Record Dates: First submitted 2020-02-10; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Pulp Disease, Dental; Dental Caries
MeSH Terms: conditions — Dental Pulp Diseases; Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioactive Glass (Experimental): 18 teeth were capped indirectly with dental adhesive containing bioactive glass applied according to the manufacturer's instructions and cured for 20 seconds and then resin composite restoration containing bioactive glass applied by golden plated composite applicator in increments 2 mm each and cured for 40 seconds for each increment.
  Interventions: Other: Bioactive Glass
- Light cured calcium hydroxide (Active Comparator): 18 teeth were capped indirectly with light cured calcium hydroxide (control group) applied according to the manufacturer's instructions by calcium hydroxide applicator and light cured for 20 seconds then resin composite restoration was applied by golden plated composite applicator in increments 2 mm each and cured for 40 seconds for each increment.
  Interventions: Other: Light cured calcium hydroxide

INTERVENTIONS:
Other: Bioactive Glass — Bioactive glass was incorporated in resin composite and its adhesive
  Arms: Bioactive Glass
Other: Light cured calcium hydroxide — Light cured calcium hydroxide
  Arms: Light cured calcium hydroxide

SUMMARY:
The aim of this study is to evaluate the effect of application of bioactive glass in different protocols on the formation of dentin bridge after indirect pulp capping using resin composite with its adhesive both are containing bioactive glass.

ELIGIBILITY:
Inclusion Criteria:

* Active carious lesion in deep dentin of molars.
* Absence of cavitated lesions at the buccal or lingual surfaces as determined by clinical and radiographic examination.
* Absence of clinical diagnosis of pulp exposure, fistula, swelling of periodontal tissues, and abnormal tooth mobility;
* Absence of clinical symptoms of irreversible pulpitis, such as spontaneous pain or sensitivity to pressure;
* The extension of the carious lesion should be such that complete caries removal would risk pulp exposure, as determined by clinical and radiographic assessment;
* Absence of radiolucencies at the interradicular or periapical regions, or thickening of the periodontal spaces, that would indicate the presence of irreversible pulp pathologies or necrosis;
* Absence of internal or external root resorption.
* Co-operative patients approving the trial.

Exclusion Criteria:

* Patients with systemic medical conditions
* pregnant females
* Teeth with spontaneous pain or sensitivity to percussion.
* Teeth with periodontal lesions, internal or external root resorption, mobility of tooth, sinus opening, or abscessed tooth.
* Radiographic examination revealed, interrupted or broken lamina dura, widened periodontal ligament space, periapical radiolucency.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Change of dentine thickness | baseline, one month, 3 months and 6 months
  Thickness in millimeters using CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- AlAzhar University, Faculty of Dentistry for Girls, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided